CLINICAL TRIAL: NCT04666896
Title: Effectiveness of a 6-month Home-based Exercise Program for Treating Shoulder Instability in Patients With Hypermobile Ehlers-Danlos Syndrome (hEDS) or Hypermobility Spectrum Disorder (HSD): A Pilot Randomized Controlled Trial.
Brief Title: Patient-based Care Versus Standard Care for Patients With hEDS/HSD and Multidirectional Shoulder Instability
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19, this pilot study ended prematurely.
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B670201939864; BOF17/DOC/220 (Other Grant/Funding Number: Bijzonder Onderzoeksfonds (BOF))
Record Dates: First submitted 2020-12-08; First posted 2020-12-14 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Hypermobile Ehlers-Danlos Syndrome; Hypermobility Syndrome; Multidirectional Subluxation of Shoulder
Keywords: Hypermobile Ehlers-Danlos syndrome; Hypermobility Spectrum Disorder; Mutlidirectional shoulder instability; Telerehabilitation
MeSH Terms: conditions — Ehlers-Danlos syndrome type 3

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evidence-based tailored care (group A) (Experimental): Patients who were randomized to group A received a tailored exercise program, with exercises developed based on recent hEDS/HSD research data.
  Interventions: Other: Tailored home-based exercise therapy
- Evidence-based standard care (group B) (Active Comparator): This exercise program was composed in order to reflect evidence-based standard care, in a telerehabilitation format.
  Interventions: Other: Standard home-based exercise therapy

INTERVENTIONS:
Other: Tailored home-based exercise therapy — exercises were divided into four types: 1) shrug exercises; 2) external rotation exercises; 3) bench slides; and 4) wall slides.
  Arms: Evidence-based tailored care (group A)
Other: Standard home-based exercise therapy — The exercise program consisted of 4 types of exercises for training 1) balance and proprioception; 2) isometric strength; 3) rotator cuff muscles; and 4) open chain elevation
  Arms: Evidence-based standard care (group B)

SUMMARY:
For hEDS or HSD patients with MDI, a multidisciplinary treatment approach is suggested. As follows, physiotherapy plays a key role in this integrative management. Nevertheless, knowledge regarding EDS is limited among health care professionals. Consequently, evidence-based treatment approaches for the hEDS/HSD population are scarce. Therefore, the aim of this study is to compare two different home-based exercise programs in order to increase our knowledge regarding treatment options, and to gain insight in safe, effective exercises for the unstable shoulder in this study population.

DETAILED DESCRIPTION:
The main purpose of this study was to evaluate the value of two telerehabilitation exercise programs for treating multidirectional shoulder instability (MDI) in patients diagnosed with the hypermobile type of The Ehlers-Danlos syndrome (hEDS) or Hypermobility Spectrum Disorders (HSD). Patients were randomly assigned to either the control group (B: evidence-based tailored care) or the experimental group (A: evidence-based standard care). Both groups received a home-based exercise program of 24 weeks. The primary outcome measure was the Western Ontario Shoulder Index (WOSI). Secondary outcomes included the Disabilities of the Arm, Shoulder and Hand (DASH), Tampa Scale for Kinesiophobia (TSK), Patient-Specific Functional Scale (PSFS), Global Rating of Change (GROC), and pain pressure thresholds (PPTs). Outcomes were assessed at baseline, after 6 weeks, 12 weeks, and at the end of the study (24 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-65 years
* Patients diagnosed by a medical doctor with generalized HSD or hEDS, according to the diagnostic criteria for hEDS and HSD as stated in the recently published international classification for the Ehlers-Danlos syndromes
* Patients diagnosed with multidirctional shoulder instability (MDI): The diagnosis of MDI was confirmed when 1) patients reported symptoms of shoulder instability in daily life (e.g. recurrent subluxations) without a traumatic onset; 2) patients scored positive on shoulder laxity and instability tests (i.e. sulcus sign, anterior and posterior load and shift, posterior jerk, Gagey hyperabduction test, passive and active external rotation in supine, apprehension and relocation test) in at least two directions; 3) patients had shoulder pain for at least three months prior to the study.

Exclusion Criteria:

* pregnancy during study participation
* patients who started a new physiotherapeutic treatment in the 2 weeks prior to the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender 'female' on ID (passport)
Enrollment: 21 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
Change in Western Ontario Shoulder Instability Index (WOSI) | Measured at baseline, 6 weeks, 12 weeks and 24 weeks, in order to assess the change in WOSI from baseline to 6 weeks, 12 weeks, and 24 weeks
  The WOSI is a responsive patient-reported and disease-specific tool, designed to be used as the primary outcome measure in clinical trials that assess treatments for patients with shoulder instability. Range 0 - 2100 points. Higher scores express worse status.

SECONDARY OUTCOMES:
The Disabilities of the Arm Shoulder and Hand (DASH) | Measured at baseline, 6 weeks, 12 weeks and 24 weeks
  The DASH is a region-specific questionnaire of upper extremity disability (range 0-100). Higher scores express worse status
The Tampa Scale for Kinesiophobia (TSK) | Measured at baseline, 6 weeks, 12 weeks and 24 weeks
  The TSK is one of the most frequently used measures for evaluating general pain-related fear of movement. Range 17 - 68 points. Higher scores express worse status.
The Patient-Specific Functional Scale (PSFS) | Measured at baseline, 6 weeks, 12 weeks and 24 weeks
  The PSFS is a patient-rated outcome measure designed to evaluate functional change. Patients were asked to identify 3 activities they were having difficulty with as a result of their shoulder instability, and to rate each activity on an 11-point Likert scale (0 = impossible to perform the activity; 10 = able to perform the activity without complaints or help). At each follow-up moment, the same 3 activities were rated. The total PSFS score was calculated by adding the scores for the 3 activities. Range 0-30 points. Higher scores express better status.
The Global Rating of Change (GROC) | Measured at baseline, 6 weeks, 12 weeks and 24 weeks
  The GROC is a transitional scale used to quantify patient-perceived improvement. It can be used to assess the results of treatment since it defines the change in health status as perceived by the patient. We asked patients to rate whether or how much their shoulder has changed since the beginning of the study on a 11 point numerical scale ('How would you describe the change in your shoulder since the beginning of the treatment program?' with -5= a lot worse; 0 = unchanged; +5= fully recovered). Range -5 to 5 points. Higher scores express better status.
Pain pressure thresholds (PPT) | Measured at baseline, 6 weeks, 12 weeks and 24 weeks
  PPTs were measured on five locations around the shoulder (local PPTs). Additionally, a distal PPT was measured at the midpoint of the quadriceps muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Fransiska Malfait, Prof. Dr., Principal Investigator — Centre of Medical Genetics
Locations (1):
- Ghent University, department of rehabilitation sciences, Ghent, Oost-Vlaanderen, Belgium